CLINICAL TRIAL: NCT01013350
Title: Prospective Observational Long-term Safety Registry of Multiple Sclerosis Patients Who Have Participated in Cladribine Clinical Studies (PREMIERE)
Brief Title: Prospective Observational Long-term Safety Registry of Multiple Sclerosis Participants Who Have Participated in Cladribine Clinical Trials
Acronym: PREMIERE
Status: Completed | Type: Observational
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR700568-012; 2009-017978-21 (EudraCT Number)
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cladribine; PREMIERE; Observational study
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Never Exposed to Cladribine: All participants who received placebo matched to cladribine in previously conducted clinical trials (NCT Number: NCT00213135, NCT00436826 , NCT00641537, NCT00938366 and NCT00725985).
- Exposed to Cladribine: All participants who received cladribine in previously conducted clinical trials (NCT Number: NCT00213135, NCT00436826, NCT00641537, NCT00938366 and NCT00725985).

SUMMARY:
Prospective Observational Long-term Safety Registry of Multiple Sclerosis Participants who Have Participated in Cladribine Clinical Trials

ELIGIBILITY:
Inclusion Criteria:

* Prior enrollment into selected oral cladribine clinical trials as of randomization to either study drug or placebo, once participation in the clinical trial has ended
* Written informed consent was given

Exclusion Criteria:

* Participants who cannot be reached by telephone
* Participants unable to answer the registry questionnaires and who do not have a next of kin or caregiver able to answer the registry questionnaires
* Participants who - either during the lag interval or subsequently enter an interventional study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with Multiple Sclerosis and had already participated in Sponsor oral cladribine clinical development trials
Sampling Method: Non-Probability Sample
Enrollment: 1161 (Actual)
Dates: Start 2009-11-30 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Outcome Sciences, Inc, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Giovannoni G, Galazka A, Schick R, Leist T, Comi G, Montalban X, Damian D, Dangond F, Cook S. Pregnancy Outcomes During the Clinical Development Program of Cladribine in Multiple Sclerosis: An Integrated Analysis of Safety. Drug Saf. 2020 Jul;43(7):635-643. doi: 10.1007/s40264-020-00948-x. PMID 32447743

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study enrolled participants from previous clinical trials (NCT00213135, NCT00436826, NCT00641537, NCT00938366 and NCT00725985) and were exposed either to placebo matched to cladribine or cladribine itself. 13 enrolled participants from NCT00938366 were excluded from safety analysis as the dose was relatively lower compared with other studies.
Period: Overall Study
Arm/Group | Never Exposed to Cladribine | Exposed to Cladribine
Started | 198 | 963
Safety Analysis Set | 198 | 950
Completed | 160 | 771
Not Completed | 38 | 192
Not completed — Lost to Follow-up | 15 | 95
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 4 | 20
Not completed — Withdrawal by Subject | 15 | 38
Not completed — Death | 3 | 5
Not completed — Participant entered interventional study | 0 | 8
Not completed — Other | 1 | 25

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants in the current study who either received placebo matched to cladribine or cladribine in previously conducted clinical trials (NCT Number: NCT00213135, NCT00436826 , NCT00641537 and NCT00725985).
Groups:
- Never Exposed to Cladribine: All participants who received placebo matched to cladribine in previously conducted clinical trials (NCT Number: NCT00213135, NCT00436826, NCT00641537 and NCT00725985).
- Exposed to Cladribine: All participants who received cladribine in previously conducted clinical trials (NCT Number: NCT00213135, NCT00436826, NCT00641537 and NCT00725985).
- Total: Total of all reporting groups
Arm/Group | Never Exposed to Cladribine | Exposed to Cladribine | Total
Number analyzed (Participants) | 198 | 950 | 1148
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (10.2) | 40.6 (10.8) | 40.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 632 | 773
  Male | 57 | 318 | 375
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 13 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 7 | 7
  White | 190 | 925 | 1115
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Drug Reactions (SADRs)
Description: SADR is an adverse drug reaction that fulfils at least one of the seriousness criterion; results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is otherwise considered as medically important. An adverse drug reaction (ADR) is a response to a medicinal product which is noxious and unintended, and which occurs at doses normally used in man for prophylaxis, diagnosis, or therapy of disease or for the restoration, correction, or modification or physiological functions. Number of participants with SADRs were reported.
Time Frame: up to 3251 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Never Exposed to Cladribine | Exposed to Cladribine
Number analyzed (Participants) | 198 | 950
Participants | 1 | 14

2. Primary Outcome: Time to Resolution of Lymphopenia, Among Registry Participants With Persistent Lymphopenia
Description: Persistent lymphopenia was defined as Grade 3 (less than [<] 500-200 per millimeter [mm] ^3 or < 0.5-0.2 multiply [*]10^9 per Liter) or Grade 4 (< 200/mm^3 or < 0.2*10^9 per Liter) lymphopenia as defined by the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. The resolution is the achievement of a CTCAE Grade 1 (< lower limit of normal [LLN] to 800 per mm^3 or < LLN to 0.8*10^9 per Liter) or Grade 0 (< 910 per mm^3 ) lymphocyte count. Persistent Lymphopenia was reported only in Cladribine group, hence results are reported only for "Exposed to Cladribine" arm. Time to resolution is reported.
Time Frame: up to 3251 days
Population: Lymphocyte Population included participants from safety analysis set who had persistent lymphopenia. Here, "overall number of participants analyzed" signified participants with resolved lymphopenia.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Exposed to Cladribine
Number analyzed (Participants) | 41
months | 30.22 (17.78)

3. Primary Outcome: Number of Participants With Adverse Events (AEs) in the "Blood and Lymphatic System Disorders" System Organ Class (SOC) and in the "Neoplasms Benign, Malignant, and Unspecified" SOC
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug.
Time Frame: up to 3251 days
Population: Safety analysis set included all participants in the current study who either received placebo matched to cladribine or cladribine in previously conducted clinical trials (NCT Number: NCT00213135, NCT00436826 , NCT00641537, NCT00725985).
Measure: Count of Participants; unit: Participants
Arm/Group | Never Exposed to Cladribine | Exposed to Cladribine
Number analyzed (Participants) | 198 | 950
Participants
  Blood and Lymphatic System Disorders SOC | 18 | 92
  Neoplasms Benign, Malignant, and Unspecified SOC | 4 | 25

4. Secondary Outcome: Number of Participants With Pregnancy Outcomes
Description: Pregnancies occurred among female participants exposed to cladribine were identified by a participant-reported positive pregnancy test and at least a 2-week delay in menses, or a participant-reported pregnancy diagnosed by a physician. Pregnancy outcomes were Live birth, Induced abortion (Termination), Spontaneous loss (Miscarriage) (< 22 weeks), Foetal death (stillbirth) (>=22 weeks), Ectopic pregnancy, Congenital malformations and others (unknown). Number of participants as per pregnancy outcome category were reported.
Time Frame: up to 3251 days
Population: Safety analysis set. Here, "Overall Number of Participants Analyzed" signifies number of participants with pregnancies.
Measure: Count of Participants; unit: Participants
Arm/Group | Never Exposed to Cladribine | Exposed to Cladribine
Number analyzed (Participants) | 34 | 57
Participants
  Live Birth | 23 | 39
  Induced Abortion (Termination) | 3 | 3
  Spontaneous Loss (Miscarriage) | 2 | 3
  Foetal Death (Still birth) | 0 | 1
  Ectopic Pregnancy | 0 | 1
  Congenital Malformations | 0 | 0
  Unknown | 6 | 10

ADVERSE EVENTS:
Time Frame: up to 3251 days
Description: Safety analysis set included all participants in the current study who either received placebo matched to cladribine or cladribine in previously conducted clinical trials (NCT Number: NCT00213135, NCT00436826, NCT00641537 and NCT00725985).
Arm/Group | Never Exposed to Cladribine | Exposed to Cladribine
All-Cause Mortality (participants affected / at risk) | 3/198 | 5/950
Serious Adverse Events (participants affected / at risk) | 10/198 | 63/950
Other Adverse Events (participants affected / at risk) | 26/198 | 124/950
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Never Exposed to Cladribine (N=198) | Exposed to Cladribine (N=950)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Dandy-Walker syndrome (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal melanosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Accidental death (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Meningoencephalitis herpetic (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Nonkeratinising carcinoma of nasopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cerebellar syndrome (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Hemiparaesthesia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 8
Optic neuritis (Nervous system disorders) | 1 | 1
Relapsing-remitting multiple sclerosis (Nervous system disorders) | 0 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Jealous delusion (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Neonatal anoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 1 | 0
Stem cell transplant (Surgical and medical procedures) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Never Exposed to Cladribine (N=198) | Exposed to Cladribine (N=950)
Lymphopenia (Blood and lymphatic system disorders) | 15 | 76
Multiple sclerosis relapse (Nervous system disorders) | 11 | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT01013350/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT01013350/SAP_001.pdf